CLINICAL TRIAL: NCT07376226
Title: Effects of Whole Fruit on Glycemic Control, Liver Fat, and Cardiovascular Disease Risk Factors in Adults With Type 2 Diabetes
Brief Title: Effects of Whole Fruit on Blood Sugar in People With Type 2 Diabetes
Acronym: FRUIT2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Courtney Peterson, Associate Professor, Department of Nutrition, Harvard School of Public Health (HSPH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-1444
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; whole fruit; dietary intervention; glycemic control; liver fat; continuous glucose monitoring; blood sugar; nutrition; fruit; glucose; insulin; blood pressure; carbohydrates; high-carbohydrate diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fatty Liver; Insulin Resistance

STUDY DESIGN:
Masking Description: Nurses and technicians who perform the assays and assessments will be blinded and will not be affiliated with the study. Data will be cleaned blinded by randomizing the order of the timepoints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole Fruit (Experimental): Participants will consume a large amount of whole fruit, constituting 50% of total calories.
  Interventions: Other: Whole Fruit

INTERVENTIONS:
Other: Whole Fruit — Participants will consume a large amount of whole fruit for 17 weeks. During the first 6.5 weeks, participants will gradually increase the amount of whole fruit they eat by 5% every 5 days. Once they reach 50% of their calories as whole fruit, they will continue to eat 50% fruit for the remaining 10.5 weeks of the study. This is a controlled feeding study, so participants will consume fruit prepared in a metabolic kitchen. The fruit will consist of fresh fruit, dried fruit, and frozen fruit blended into smoothies. To demonstrate compliance, participants will video-record themselves eating the provided fruit. All participants will receive the same dietary intervention. Participants will otherwise continue their usual diet and lifestyle habits.

SUMMARY:
This study will determine the effects of consuming whole fruit on blood sugar control, liver fat, and cardiovascular health in adults with type 2 diabetes who are not treated with insulin.

DETAILED DESCRIPTION:
Diabetes is one of the top three drivers of healthcare costs in the U.S., and nearly half of Americans will develop either diabetes or prediabetes in their lifetime. It is therefore critical to find new strategies to treat or reverse diabetes.

One such approach is adopting a healthy diet, which can dramatically improve blood sugar levels in adults with type 2 diabetes and even induce diabetes remission in some patients. Despite this, not much is known about which food groups are most effective at improving blood sugar levels in patients with diabetes.

Although individuals with type 2 diabetes are often advised to reduce carbohydrate intake, current dietary guidelines also recommend consuming fruit and other carbohydrate-rich foods. This has led to confusion among patients and clinicians about whether eating fruit, particularly in larger amounts, is beneficial or harmful for blood sugar and overall health. Whole fruit differs from many other carbohydrate sources in that whole fruit is rich in fiber, vitamins, minerals, and bioactive plant compounds, while being relatively low in energy density.

Most prior research examining the effects of whole fruit in people with type 2 diabetes has been epidemiologic, focused on individual fruits, or combined whole fruit with fruit juice and/or vegetables into a single food category. As a result, it is unknown how whole fruit, as a food category, affects glycemic control and cardiovascular health.

The investigators previously found that a whole-fruit-rich, Mediterranean-style diet improved blood sugar control and blood pressure in patients with type 2 diabetes and even allowed some patients to wean off all anti-hyperglycemic medications. The investigators will conduct a follow-up study to determine the effects of whole fruit alone on glycemic control, liver fat, and cardiovascular risk factors. The study will be a single-arm controlled feeding study to determine the effects of eating a large amount of whole fruit for 17 weeks on glycemic control (Aim 1), liver fat (Aim 2a), and cardiovascular disease risk factors (Aim 2b) in patients with insulin-independent type 2 diabetes. The primary measures of glycemic control will be mean 24-hour glucose levels (as measured by continuous glucose monitoring) and mean 3-hour glucose levels (as measured during a 3-hour oral glucose tolerance test). These assessments will be supplemented by, and interpreted in light of, other glycemic outcomes, which are listed as outcomes #3-9 below.

By providing controlled, high-quality evidence, this study will determine whether whole fruit is good or bad for patients with type 2 diabetes and will improve dietary guidelines for the hundreds of millions of individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Diagnosed with type 2 diabetes
* HbA1c between 6.5-12.0%
* Fasting C-peptide level ≥0.5 ng/ml, indicating the patient does not have beta-cell failure, as measured at screening

Exclusion Criteria:

* On insulin
* Evidence of latent autoimmune diabetes (LADA) or maturity-onset diabetes of the young (MODY)
* Estimated glomerular filtration rate (eGFR) <45 ml/min per 1.73 m²
* Heart attack in the past 6 months or severe/unstable heart failure
* On weight loss medication, including GLP-1 receptor agonists (e.g., semaglutide, dulaglutide)
* Change in the dosage of a chronic medication that may affect study endpoints within the past 3 months
* Clinically significant laboratory abnormality (e.g., abnormal hemoglobin levels)
* Significant gastrointestinal disease, major gastrointestinal surgery, or gallstones
* Significant cardiovascular, renal, cardiac, liver, lung, adrenal, or nervous system disease that might compromise participant safety or data validity
* Evidence of cancer (other than non-melanoma skin cancer) within the last 5 years
* Lost or gained more than 5 lbs (or more than 2% of body weight if the patient weighs >250 lbs) of weight in the past 2 months
* Pregnant, planning to become pregnant in the next 6 months, or breastfeeding
* Major psychiatric condition that would affect the ability to participate in the study
* Not able to eat the provided study meals (e.g., food allergies)
* Behavioral factors or circumstances that may impede adherence to the dietary intervention
* Not able to undergo the MRI scan (e.g., due to claustrophobia, implanted metal objects, or body girth ≥60 cm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Mean 24-hour Glucose Levels | Change from baseline to week 17
  Average 24-hour interstitial glucose levels (mg/dl), as measured by continuous glucose monitoring (CGM). If needed, data will be adjusted for any changes in antihyperglycemic medication use, using the medication effect score (MES).
Mean 3-hour Glucose Levels | Change from baseline to week 17
  Mean glucose (mg/dl) during a 3-hour oral glucose tolerance test (OGTT)
Mean 3-hour Insulin | Change from baseline to week 17
  Mean insulin (mU/l) during a 3-hour OGTT
Mean 3-hour C-Peptide | Change from baseline to week 17
  Mean C-Peptide (ng/ml) during a 3-hour OGTT
Insulin Sensitivity | Change from baseline to week 17
  Insulin sensitivity (dl/kg/min/μU/ml) during a 3-hour OGTT, as measured by the Oral C-Peptide Minimal Model
Dynamic Beta-Cell Responsivity | Change from baseline to week 17
  Phi_dynamic during a 3-hour OGTT, as measured by the Oral C-Peptide Minimal Model (which is a set of 5 coupled differential equations; see reference under Citations). Phi_dynamic is a measure of beta-cell responsiveness during first-phase insulin secretion. It is a dimensionless index (arbitrary units), where higher values denote greater insulin secretion
Static Beta-Cell Responsivity | Change from baseline to week 17
  Phi_static during a 3-hour OGTT, as measured by the Oral C-Peptide Minimal Model (which is a set of 5 coupled differential equations; see reference under Citations). Phi_static is a measure of beta-cell responsiveness during second-phase insulin secretion. The units of measure are min^-1, and higher values denote greater insulin secretion.
Glycemic Variability | Change from baseline to week 17
  Measures of glucose variability derived from continuous glucose monitoring, including mean amplitude of glycemic excursions and standard deviation (mg/dl).
Time-in-range Metrics from CGM | Change from baseline to week 17
  Standard time-in-range metrics, including time-below-range (TBR), time-in-range (TIR), and time-above-range (TAR), as standardized by the International Consensus on Time in Range. Values will be reported as percentages of the 24-hour day.

SECONDARY OUTCOMES:
Intrahepatic Lipid (Liver Fat) | Change from baseline to week 17
  Percentage as measured using Magnetic Resonance Spectroscopy (MRS) and 3-point M-Dixon Magnetic Resonance Imaging (MRI)
Body Weight | Change from baseline to week 17
  kg
Systolic and Diastolic Blood Pressure | Change from baseline to week 17
  mm Hg
Heart Rate | Change from baseline to week 17
  beats per minute
Lipids | Change from baseline to week 17
  Fasting total cholesterol (mg/dl), LDL cholesterol (mg/dl), HDL cholesterol (mg/dl), and triglycerides (mg/dl).

CONTACTS AND LOCATIONS:
Overall Officials: Courtney M Peterson, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard T. H. Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cobelli C, Dalla Man C, Toffolo G, Basu R, Vella A, Rizza R. The oral minimal model method. Diabetes. 2014 Apr;63(4):1203-13. doi: 10.2337/db13-1198. PMID 24651807